CLINICAL TRIAL: NCT07365280
Title: An Open-Label, Multicenter, Randomized Phase II Study to Evaluate the Efficacy and Safety of Personalized Dendritic Cell Vaccine ZSNeo-DC1.1 in Combination With Temozolomide as Adjuvant Therapy in Patients With Newly Diagnosed Glioblastoma After Surgery and Concurrent Chemoradiotherapy
Brief Title: Neoantigen-Pulsed Autologous Dendritic Cell Vaccine Combined With Temozolomide for Newly Diagnosed Glioblastoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ZSky Biotech Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSKY2025-1005
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: DC; Personalized neoantigen-pulsed autologous dendritic cells vaccine
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Personalized dendritic cell vaccine ZSNneo-DC1.1 in combination with temozolomide.
  Interventions: Biological: Personalized Dendritic Cell Vaccine ZSNeo-DC1.1; Drug: Temozolomide (TMZ)
- Control (Active Comparator): Standard adjuvant temozolomide chemotherapy alone
  Interventions: Drug: Temozolomide (TMZ)

INTERVENTIONS:
Biological: Personalized Dendritic Cell Vaccine ZSNeo-DC1.1 — Patients receive six subcutaneous injections of ZSNeo-DC1.1 during adjuvant temozolomide chemotherapy. ZSNeo-DC1.1 is administered at a fixed dose of 1 × 10⁷ cells per injection according to the assigned immunization schedule. Temozolomide is administered as per protocol.
  Other Names: Temozolomide
  Arms: Experimental
Drug: Temozolomide (TMZ) — Patients receive standard adjuvant temozolomide chemotherapy alone

SUMMARY:
This is a multicenter, open-label, randomized Phase II clinical study designed to evaluate the efficacy and safety of a personalized dendritic cell (DC) vaccine, ZSNeo-DC1.1, in combination with temozolomide (TMZ) as adjuvant therapy in patients with newly diagnosed glioblastoma (GBM).

Eligible patients with histologically confirmed, IDH1/IDH2 wild-type newly diagnosed glioblastoma who have undergone tumor debulking surgery followed by standard concurrent chemoradiotherapy will be enrolled. After confirmation of tumor neoantigens and eligibility, patients will be randomized in a 1:1 ratio to receive either ZSNeo-DC1.1 in combination with TMZ or TMZ alone.

The primary objective is to evaluate progression-free survival (PFS) as assessed by an Independent Radiological Review Committee (IRRC) according to RANO 2.0 criteria. Secondary objectives include overall survival (OS), survival rates, tumor response outcomes, and safety. Exploratory objectives include assessment of antigen-specific T-cell immune responses induced by ZSNeo-DC1.1.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible:

Inclusion Criteria

1. Age 18 to 75 years, inclusive
2. Histologically confirmed newly diagnosed glioblastoma (WHO grade IV)
3. Molecular diagnosis of IDH1/IDH2 wild-type
4. Completion of tumor debulking surgery followed by standard concurrent chemoradiotherapy
5. Karnofsky Performance Status (KPS) score of 50 to 100
6. Adequate hematologic, hepatic, renal, and coagulation function
7. Availability of sufficient tumor tissue and blood samples for neoantigen identification
8. Adequate venous access for PBMC collection
9. Life expectancy greater than 3 months
10. Willingness to use effective contraception during study treatment and for 3 months thereafter
11. Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

Exclusion Criteria:

Subjects meeting any of the following criteria are ineligible:

1. Not suitable for standard temozolomide-based chemoradiotherapy
2. Prior participation in another interventional clinical trial within 4 weeks before randomization
3. Prior implantation of carmustine wafers within 6 months
4. Known hypersensitivity to temozolomide or dacarbazine
5. Active autoimmune disease or requirement for systemic immunosuppressive therapy
6. Active infection including HIV, active hepatitis B or C, or syphilis
7. Use of systemic immunosuppressive therapy within 30 days before randomization
8. Uncontrolled cardiovascular, metabolic, or systemic disease
9. Pregnancy or breastfeeding
10. Any condition that, in the investigator's judgment, would interfere with study participation or interpretation of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2028-12-24 (Estimated); Study Completion 2028-12-24 (Estimated)

PRIMARY OUTCOMES:
PFS | From randomization until disease progression or death, whichever occurs first，assessed up to 24 months
  Progression-free survival assessed by an Independent Radiological Review Committee according to RANO 2.0 criteria

SECONDARY OUTCOMES:
OS | From randomization until death from any cause，assessed up to 36 months
  From randomization until death from any cause
Overall Survival Rates | 12 months, 18 months, and 24 months
Investigator-Assessed Progression-Free Survival | From randomization until disease progression or death，assessed up to 24 months
Disease Control Rate (DCR) | During treatment period
Best Overall Response (BOR) | During treatment period
6. Clinical Benefit Rate (CBR) | During treatment period
Safety and Tolerability | From first dose until 30 days after last dose，assessed up to 24 months
  Incidence and severity of adverse events and serious adverse events graded according to NCI CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No